CLINICAL TRIAL: NCT04161690
Title: Evaluation of Dexketoprofen Given Intravenous or Intrathecal in Postoperative Pain in Patients Undergoing Total Knee Arthroplasty
Brief Title: Evaluation of Dexketoprofen in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Elena Nikolakopoulou, Principal Investigator, KAT General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13022
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — dexketoprofen trometamol; Ropivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group IV (Active Comparator): Dexketoprofen 50mg is given intravenous 10 min before the start of the surgery. Local infiltration analgesia is proceeded by the surgeon with 300mg ropivacaine.
  Interventions: Drug: Dexketoprofen Trometamol; Drug: Ropivacaine Hydrochloride 7.5 MG/ML
- Group Periarticular (Active Comparator): Dexketoprofen 50mg is given as part of the local infiltration analgesia with 300mg ropivacaine. Local infiltration analgesia is proceeded by the orthopedic surgeon.
  Interventions: Drug: Dexketoprofen Trometamol; Drug: Ropivacaine Hydrochloride 7.5 MG/ML
- Group P (Placebo Comparator): Local infiltration analgesia is proceeded by the surgeon with 300mg ropivacaine.
  Interventions: Drug: Ropivacaine Hydrochloride 7.5 MG/ML

INTERVENTIONS:
Drug: Dexketoprofen Trometamol — intravenous dexketoprofen 50mg or intrathecal
  Arms: Group IV; Group Periarticular
Drug: Ropivacaine Hydrochloride 7.5 MG/ML — Local Infiltration Analgesia

SUMMARY:
Pain is a global public health issue and represents the most common reason for both physician consultation and hospital admissions. Dexketoprofen is a new NSAID treating acute postoperative pain. The purpose of this study is to evaluate the analgesic effect when it is given intravenously or as part of the local infiltration analgesia in patients under spinal anesthesia undergoing unilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* unilateral total knee arthroplasty
* accept to enter the study
* ASA score I or II
* hospitalization for at least 2 days

Exclusion Criteria:

* allergy in any given medications
* active gastrointestinal bleeding or other active bleeding
* history of peptic ulcer
* renal failure
* hepatic failure
* chronic heart failure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
VAS Score in 8hours after surgery | 8h
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. 10 describes the worst pain that a person ever imagined.
VAS Score 24hours after surgery | 24h
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
VAS Score 48hours after surgery | 48h
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Total tramadol consumption the first 24hours | 24h

CONTACTS AND LOCATIONS:
Locations (1):
- Elena Nikolakopoulou, Athens, Kifissia, Greece

IPD SHARING:
Plan to Share IPD: Undecided